CLINICAL TRIAL: NCT01082978
Title: A Randomized Controlled Trial of Portable Electronic(USB)and Paper Medical Records as an Adjunct to Usual Care (Portable Health File RCT): an Evaluation of Short Term Quality Measures and Long-term Clinical Outcomes
Brief Title: Portable Health Files Improve Quality of Care and Health Outcomes: a Randomized Controlled Trial
Acronym: PHF-RCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: St George Hospital, Australia (Other)
Collaborators: South Eastern Area Health Service (Other); The University of New South Wales (Other); National Health and Medical Research Council, Australia (Other)
Responsible Party: Principal Investigator, Marissa Lassere, Senior Staff Specialist, St George Hospital, Australia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: PHF-06-124-ML; NHMRC 455467 (Other Grant/Funding Number: NHMRC)
Record Dates: First submitted 2010-03-08; First posted 2010-03-09 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Chronic Medical Conditions; Personal Health Records; Electronic Medical Record
Keywords: Quality of Life; Health Care Quality and Safety; Randomized controlled trial

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Primary outcomes, death and overnight hospitalisations, are obtained through record linkage and are masked outcomes. Outcome assessor, however, is not masked to patient-reported outcomes. Chief Investigator and statistical analyses are masked to randomisation/intervention group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No

ARMS (3):
- Electronic (USB) Portable Health File (Experimental): Patients randomized to this arm of the trial will be given a USB memory device that contains the Portable Health File (PHF) software. The portable health files contained core medical data which functions as a subset of a comprehensive medical record. The portable health file is updated by the health care provider at each visit and could also be updated by patient between visits if necessary.
  Interventions: Device: Electronic (USB) Portable Health File
- Paper Portable Health File (Experimental): Patients randomized to this arm of the trial will be given the paper Portable Health File. The paper Portable Health File contains core medical and other important data which functions as a subset of a more comprehensive medical record. This paper-based portable health file is updated by health care providers at each visit. The PHF can also be updated by patient between visits.
  Interventions: Device: Paper Portable Health File
- Usual standard of care (No Intervention): Patients randomized to this arm of the trial will not be given a Portable Health File. This arm is the concurrent control comparator arm.

INTERVENTIONS:
Device: Electronic (USB) Portable Health File — Patients randomized to this arm of the trial will be given a USB memory device that contains the Portable Health File (PHF) software. The portable health files contained core medical data which functions as a subset of a comprehensive medical record. The portable health file is updated by the health care provider at each visit and could also be updated by patient between visits if necessary.
  Other Names: Electronic Personal Health Record; Electronic Patient-Health Provider Shared Medical Record; Electronic Patient-Health Provider Shared Journal; Electronic Patient-carried Shared Medical Record; Electronic Patient-carried Continuity of Care Record
  Arms: Electronic (USB) Portable Health File
Device: Paper Portable Health File — Patients randomized to this arm of the trial will be given the paper Portable Health File. The paper Portable Health File contains core medical and other important data which functions as a subset of a more comprehensive medical record. This paper-based portable health file is updated by health care providers at each visit. The PHF can also be updated by patient between visits.
  Other Names: Paper Personal Health Record; Paper Patient-Health Provider Shared Medical Record; Paper Patient-Health Provider Shared Journal; Paper Patient-carried Shared Medical Record; Paper Patient-carried Continuity of Care Record
  Arms: Paper Portable Health File

SUMMARY:
The PHF trial will assess the acceptability and long term outcomes resulting from the usage of electronic (carried by the patient on a USB memory device) and paper portable health files in a population with high intensity use of medical services. The rationale is that use of the portable health files provides a conduit of direct communication among health care providers of a patient's important health care information and this leads to better care and patient outcomes.

Primary hypothesis: Addition of a patient-held portable health file (PHF) to usual care improves patient outcome and quality-of-life compared to usual care alone.

Secondary hypothesis: Addition of patient-held portable health file (PHF) to usual care is acceptable and satisfactory to patients and their health care providers.

DETAILED DESCRIPTION:
A common problem faced by patients and clinicians in our health system is continuity of care and 'clinical handovers'. Few medical record technologies, paper or electronic, top down or bottom up, have been evaluated in a randomised clinical outcome trial to determine the clinical benefits and costs of 'shared' medical and health information. Furthermore, although there are many studies that have evaluated processes of care only a minority do so within a randomized design. Given that any difference is, possibly, small to moderate in magnitude, and given confounders, the use of a randomisation is an essential design requirement.

The first 12 months of the trial constitutes Stage 1 whose primary objective is to describe the acceptability and satisfaction of the our Portable Health Files, and other key process measures. The subsequent 36 months constitutes Stage 2 whose primary objective it to compare important clinical outcomes. The assigned treatment (i.e., the e-PHF or p-PHF) will be used for 4 years total.

To take into account a probable lag effect of the interventions, patients will also be followed for an additional 3 years beyond the conclusion of the randomised trial to see if there are any longer-term effects.

The trial is un-blinded so there will be a potential for bias in trial conduct and a potential for ascertainment bias in the determination of important clinical outcomes and quality-of-life. To reduce clinical outcome ascertainment bias a blinded Adjudication Committee will make the determination which out-of-hospital events are "serious". The other primary outcomes: mortality and all overnight hospitalizations are objective outcomes and are not subject to ascertainment bias.

Secondary outcomes include quality of life, quality measures uptake, investigations, medication use, medication errors, and adverse drug reactions. Utilities and costs will also be collected for cost-effectiveness analysis. Patient and provider acceptability and satisfaction with the PHFs will be also collected.

All primary analyses will be undertaken masked to randomized arm allocation.

Most secondary analyses including quality of life, quality measures uptake, investigations, medication use, medication errors, and adverse drug reactions, health utilities, health care utilisation and health care costs will also be undertaken masked to randomized arm allocation.

This Adjudication Committee will also monitor trial safety and scientific integrity.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be of age 60 or greater
2. Patients living independently in the community. Hostel care is acceptable, but patients that are not independent requiring full nursing home care are excluded.
3. Subjects must have had six medical practitioner visits in the previous 12 months
4. Subjects must have at least two of the following confirmed chronic diseases that require prescription oral or parenteral drug treatment or surgery and requiring at least annual specialist consultation: cardiovascular, respiratory, endocrine, renal, neurologic, gastrointestinal, hepatic, genitourinary, haematologic. infective, rheumatic, inflammatory, immunologic or neoplastic disease.

6. Subject's GP must have access to a computer during the consultation visit. 7. Subjects must have at least two medical specialists at least one of whom has access to a computer during the consultation visit.

8. Subjects must be able to understand the purpose of the trial and undergo full and valid informed consent.

Exclusion Criteria:

1. Life expectancy of less than 12 months.
2. Inability to carry a paper PHF or e-PHF and having no care-giver willing and able to accomplish same.
3. Mentally unable to undertake valid informed consent.
4. Patients who are not independent in the community, that cannot mobilise to see a specialist or requiring full nursing home care

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 382 (Estimated)
Dates: Start 2010-03 (Actual); Primary Completion 2019-03 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Combined endpoint of deaths, hospitalisations (excepting day only hospitalisations), and serious out-of-hospital events | 48 months + 36 month extension
  The primary outcome is the total number of important clinical events (all hospitalisations except same-day hospitalisations, all serious out-of-hospital events and deaths).
  See above: The assigned treatment (i.e., the e-PHF or p-PHF) will be used for 4 years total. Patients will also be followed for an additional 3 years beyond the conclusion of the randomised trial to see if there are any longer-term lag effects.

SECONDARY OUTCOMES:
Quality of Life | every 12 months for 48 months
  SF-36 and EQ-5D
health service utilisation and health care costs | every 12 months for 48 months
  Emergency Department encounters, General Practitioner and Specialist Encounters via record linkage, and their estimated costs by MBS and other costs data
medication errors, duplicative investigations | every 12 months for 48 months
  Questionnaire, Self-report PROs and CROs
clinical workflow | every 6 months for 2 years then every 12 months until 48 months
  Questionnaire, Self-report PROs and CROs
subject and health care provider acceptability and satisfaction with portable health files (PHF) | every 3 months for 12 months then every 6 months 24 months then every 12 months until 48 months
  Questionnaire, Self-report PROs and CROs
guidelines uptake and documentation | every 6 months for 24 months then every 12 months until 48 months
  Questionnaire, Self-report PROs and CROs
health literacy | every 12 months until 48 months
  Questionnaire, Self-report PROs
information technology and computer expertise | every 6 months for 24 months then every 12 months until 48 months
  Questionnaire, Self-report PROs
adverse events | every 3 months for 24 months then every 6 months until 48 months
  Questionnaire, Self-report PROs

CONTACTS AND LOCATIONS:
Overall Officials: Marissa ND Lassere, MBBS PhD, Study Chair — St George Hospital and Univeristy of NSW; Kent R Johnson, MD, Principal Investigator — Newcastle University; George Rubin, MD, Principal Investigator — South East Sydney Area Health Service; Anthony Sara, MBBS MBA, Principal Investigator — South East Sydney Area Health Service; Andrew Parle, BSc (Hons) PhD, Principal Investigator — Consultant
Locations (1):
- St George Hospital, Kogarah, New South Wales, Australia

REFERENCES:
- [Derived] Lassere MN, Baker S, Parle A, Sara A, Johnson KR. Improving quality of care and long-term health outcomes through continuity of care with the use of an electronic or paper patient-held portable health file (COMMUNICATE): study protocol for a randomized controlled trial. Trials. 2015 Jun 4;16:253. doi: 10.1186/s13063-015-0760-8. PMID 26040644